CLINICAL TRIAL: NCT06953349
Title: Real-World Efficacy of Hydrus Microstent With OMNI Surgical System in Combination With Phacoemulsification: a Retrospective Analysis
Brief Title: Efficacy of Surgical Systems in Combination With Phacoemulsification: a Retrospective Analysis
Status: Recruiting | Type: Observational
Sponsor: Barnet Dulaney Perkins Eye Centers (Network)
Collaborators: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Alcon - IIT Proposal 95537309
Record Dates: First submitted 2025-03-04; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Open-Angle Glaucoma
Keywords: Hydrus Microstent; OMNI Surgical System; Phacoemulsification
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Group/Cohort retrospectively utilized: This will be 300 eyes that have undergone the combination of Phacoemulsification, OMNI Canaloplasty and Hydrus microstent that will successfully lower IOP in ethnically-diverse patients with Open Angle Glaucoma
  Interventions: Procedure: Real-World efficacy of Hydrus Microstent with OMNI Surgical System in combination with Phacoemulsification: a retrospective analysis

INTERVENTIONS:
Procedure: Real-World efficacy of Hydrus Microstent with OMNI Surgical System in combination with Phacoemulsification: a retrospective analysis — The use of combination Phacoemulsification, OMNI Canaloplasty and Hydrus microstent successfully lowers IOP in ethnically-diverse patients with Open Angle Glaucoma
  Other Names: OMNI; Hydrus Microstent

SUMMARY:
Real-World efficacy of Hydrus Microstent with OMNI Surgical System in combination with Phacoemulsification: a retrospective analysis

DETAILED DESCRIPTION:
The use of combination Phacoemulsification, OMNI Canaloplasty and Hydrus microstent successfully lowers IOP in ethnically-diverse patients with Open Angle Glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Subjects with h/o CEIOL/OMNI/Hydrus (chosen based on subjects on more than 1 medication pre-operatively) with at least 3 years of follow up data
* have Glaucoma

Exclusion Criteria:

* Patients with angle closure glaucoma or secondary forms of glaucoma due to neovascularization of the angle, uveitic glaucoma, congenital glaucoma, or glaucoma due to congenital anomalies.
* Patients with refractory CME or CME persisting 3 months or more post-operatively
* Patients with incomplete IOP, medication logs or VF data within post-operative period
* Prior incisional surgery or MIGS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 subjects that have undergone CEIOL/OMNI/Hydrus
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measured Efficacy of Surgical Process with Phacoemulsification | 24 months
  Primary endpoint stratified by complete or qualified success:
  • Proportion of patients with complete success (%) - without the use of medications

SECONDARY OUTCOMES:
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Proportion of patients with qualified success (%) - with glaucoma meds without increase from baseline
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Overall IOP reduction from baseline (mmHg)
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Overall medication reduction (#0-5)
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Rate of mean deviation change (dB)
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • SSIs (% on trabeculectomy, glaucoma drainage implant (GDI), other)
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  Additional Secondary Endpoint stratified by Complete or Qualified surgical success defined by the following:
  * Complete success: Without the use of glaucoma medications
  * Qualified success: Using glaucoma medications, but without an increase from the baseline number
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Overall medication reduction from baseline, measured at 12, 24 and 36 month timepoints
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Overall IOP reduction from baseline, measured at 12, 24 and 36 month timepoints
Additional Benefits of the Surgical System and Phacoemulsification | 36 months
  • Rate of mean deviation change from baseline to postop time points in Humphrey visual field tests

CONTACTS AND LOCATIONS:
Overall Officials: Christine Funke, Medical Doctor, Principal Investigator — Barnet Dulaney Perkins Eye Centers
Locations (1):
- Barnet Dulaney Perkins Eye Center, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
To report on surgical success after cataract surgery in ethnically diverse (Caucasian, Asian, African American, Hispanic, Tribal) patients with multiple glaucoma using combined MIGS procedures.
Supporting Information: Study Protocol, CSR
Time Frame: IPD will be made available once the study data collection is complete tentatively 12/2025 for a period of 12 months, to tentatively 12/2026
Access Criteria: The investigators will allow fellow researchers access to the data as the investigators work to publish the findings.
URL: http://goodeyes.com

REFERENCES:
- [Background] Montesano G, Ometto G, Ahmed IIK, Ramulu PY, Chang DF, Crabb DP, Gazzard G. Five-Year Visual Field Outcomes of the HORIZON Trial. Am J Ophthalmol. 2023 Jul;251:143-155. doi: 10.1016/j.ajo.2023.02.008. Epub 2023 Feb 21. PMID 36813144
- [Background] Hirsch L, Cotliar J, Vold S, Selvadurai D, Campbell A, Ferreira G, Aminlari A, Cho A, Heersink S, Hochman M, Gallardo M, Williamson B, Phan R, Nelson C, Dickerson JE Jr. Canaloplasty and trabeculotomy ab interno with the OMNI system combined with cataract surgery in open-angle glaucoma: 12-month outcomes from the ROMEO study. J Cataract Refract Surg. 2021 Jul 1;47(7):907-915. doi: 10.1097/j.jcrs.0000000000000552. PMID 33315733
- [Background] Sarkisian SR Jr, Radcliffe N, Harasymowycz P, Vold S, Patrianakos T, Zhang A, Herndon L, Brubaker J, Moster R, Francis B; ASCRS Glaucoma Clinical Committee. Visual outcomes of combined cataract surgery and minimally invasive glaucoma surgery. J Cataract Refract Surg. 2020 Oct;46(10):1422-1432. doi: 10.1097/j.jcrs.0000000000000317. PMID 32657904
- [Background] Laroche D, Desrosiers A, Ng C. Short-term report of early glaucoma surgery with a clear lens extraction and an intraocular lens, OMNI canaloplasty, and a HYDRUS microstent: a case series in younger patients. Front Ophthalmol (Lausanne). 2024 Jan 5;3:1288052. doi: 10.3389/fopht.2023.1288052. eCollection 2023. PMID 38983083
- [Background] Creagmile J, Kim WI, Scouarnec C. Hydrus Microstent implantation with OMNI Surgical System Ab interno canaloplasty for the management of open-angle glaucoma in phakic patients refractory to medical therapy. Am J Ophthalmol Case Rep. 2022 Nov 10;29:101749. doi: 10.1016/j.ajoc.2022.101749. eCollection 2023 Mar. PMID 36544749